CLINICAL TRIAL: NCT05087953
Title: Comparative Analysis of the Autonomic Profile Between Patients With Hereditary Amyloidotic Cardiomyopathy Caused by Transthyretin and Patients With Transthyretin Gene Mutation, Without Cardiomyopathy
Brief Title: Autonomic Evaluation of Patients With Hereditary Amyloidotic Cardiomyopathy: Hereditary Amyloidotic Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fleury (Unknown)
Responsible Party: Sponsor
Other Study IDs: SDC 5045/20/074
Record Dates: First submitted 2021-10-08; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Autonomic Nervous System Disease; Amyloid Neuropathies
MeSH Terms: conditions — Amyloid Neuropathies | interventions — Tilt-Table Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- FAC group: Patients with familial amyloidotic cardiomyopathy.
  Interventions: Diagnostic Test: Head-Up Tilt table test; Diagnostic Test: Heart Rate Variability
- Non-FAC group: Patients with transthyretin gene mutations who do not have FAC.
  Interventions: Diagnostic Test: Head-Up Tilt table test; Diagnostic Test: Heart Rate Variability
- Control group: Healthy subjects.
  Interventions: Diagnostic Test: Head-Up Tilt table test; Diagnostic Test: Heart Rate Variability

INTERVENTIONS:
Diagnostic Test: Head-Up Tilt table test — Autonomic response assessment in the orthostatic head up tilt test.
  Other Names: Tilt-test
Diagnostic Test: Heart Rate Variability — Assessment of heart rate variability on 24-hour Holter monitoring..

SUMMARY:
Transthyretin amyloidosis exhibits a variety of possible phenotypes, the hereditary neurological form being the most commonly found and studied (familial amyloidotic polyneuropathy or FAP), which can present from oligosymptomatic patients to patients with peripheral sensorimotor polyneuropathy of varying degrees and dysautonomia.

Although a specific mutation usually causes a specific phenotype, that is, with a predominantly cardiac or preferential neurological profile, with the increase in the number of diagnosed cases, an overlapping of clinical presentations has been observed.

The assessment of the autonomic profile in individuals with familial amyloidotic cardiomyopathy (FAC) has not been well studied, and it is not known whether patients with an exclusively cardiac profile of the disease may present dysautonomia or whether even mutation carriers without cardiac involvement may exhibit it.

In this study, the autonomic profiles of patients with familial amyloidotic heart disease will be compared with the profiles of patients who have mutations but without established heart disease and healthy individuals (control group).

ELIGIBILITY:
Inclusion Criteria:

* FAC group: patients with familial familial amyloidotic cardiomyopathy (FAC).
* Non-FAC group: patients with transthyretin gene mutations who do not have FAC.
* Control group: healthy, asymptomatic individuals without comorbidities and without transthyretin gene mutations.
* Agreement and signing the informed consent form.

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Ischemic or hemorrhagic stroke within the last 6 months;
  * History of ischemic heart disease;
  * Pregnancy;
  * Severe lung disease;
  * Resistant systemic arterial hypertension;
  * Diabetics;
  * Presence of pacemaker or CDI.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Autonomic response profile of patients with FAC. | 6 months
  To compare the autonomic profile by analyzing the heart rate variability on 24 hours Holter monitoring, the patterns of chronotropic and pressure response and the valsalva maneuver in the tilt table test of patients with FAC, with individuals with mutations of the transthyretin gene without FAC and in healthy individuals.

SECONDARY OUTCOMES:
Correlation between dysautonomia and electrophysiological cardiac disturbances. | 6 months
  Evaluate the relationship of dysautonomia with atrioventricular, intraventricular, interventricular conduction disturbances, presence of late potentials in the high-resolution electrocardiogram and occurrence of supraventricular and ventricular arrhythmias on Holter monitoring.
Correlation between dysautonomy and structural cardiac alterations. | 6 months
  Evaluate the relationship of dysautonomia changes with cardiac structural changes assessed by strain echocardiography.

CONTACTS AND LOCATIONS:
Locations (3):
- Brazil (3):
  - Instituto do Coração - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo
  - University of Sao Paulo Medical School - The Heart Institute, São Paulo
  - Fabio Fernandes, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rapezzi C, Quarta CC, Riva L, Longhi S, Gallelli I, Lorenzini M, Ciliberti P, Biagini E, Salvi F, Branzi A. Transthyretin-related amyloidoses and the heart: a clinical overview. Nat Rev Cardiol. 2010 Jul;7(7):398-408. doi: 10.1038/nrcardio.2010.67. Epub 2010 May 18. PMID 20479782
- [Background] Cruz MW. Regional differences and similarities of familial amyloidotic polyneuropathy (FAP) presentation in Brazil. Amyloid. 2012 Jun;19 Suppl 1:65-7. doi: 10.3109/13506129.2012.673183. Epub 2012 Apr 12. PMID 22494049
- [Background] Queiroz MC, Pedrosa RC, Berensztejn AC, Pereira Bde B, Nascimento EM, Duarte MM, Pereira-Junior PP, Cruz MW. Frequency of Cardiovascular Involvement in Familial Amyloidotic Polyneuropathy in Brazilian Patients. Arq Bras Cardiol. 2015 Nov;105(5):503-9. doi: 10.5935/abc.20150112. Epub 2015 Sep 8. PMID 26351985
- [Background] Cruz MW, Foguel D, Berensztejn AC, Pedrosa RC, Mundayat R, Ong ML; THAOS Investigators. The demographic, genetic, and clinical characteristics of Brazilian subjects enrolled in the Transthyretin Amyloidosis Outcomes Survey. Amyloid. 2017 Mar;24(sup1):103-104. doi: 10.1080/13506129.2017.1291423. No abstract available. PMID 28434317